CLINICAL TRIAL: NCT05233631
Title: Therapeutic Endoscopic Ultrasound (EUS) Registry
Brief Title: Therapeutic EUS Registry
Acronym: T-EUS
Status: Enrolling by invitation | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 030.GID.2019.D
Record Dates: First submitted 2021-10-27; First posted 2022-02-10 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Gastrointestinal Disease
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- T-EUS Patients: Any patient who has undergone clinically indicated and/or standard of care T-EUS procedures from October 2014 - June 2022.
  Interventions: Procedure: Therapeutic Endoscopic ultrasound

INTERVENTIONS:
Procedure: Therapeutic Endoscopic ultrasound — A minimally invasive procedure to assess digestive (gastrointestinal) and lung diseases. Procedure allows detailed imaging of the regional anatomy by approximating the frequency transducer to the region of interest.
  Other Names: T-EUS

SUMMARY:
The purpose of this prospective registry is to assess long-term data on efficacy, safety and clinical outcome of Therapeutic Endoscopic ultrasound (T-EUS) . The registry will evaluate technical feasibility, clinical outcome, safety profile and overall clinical management through medical chart review. The procedures we are evaluating are all clinically indicated and will not be prescribed to someone to participate in this research study.

DETAILED DESCRIPTION:
This study is a prospective, observational, medical chart review. There will be a retrospective chart review for patients who underwent endoscopic suturing procedures from October 2014 - May 2019. Those subjects will undergo no additional tests and procedures as part of this study.

In order to validate these procedures and broaden its use beyond tertiary centers, it is crucial to understand its efficacy and success rate. The objective of the study is to evaluate retrospectively and prospectively the efficacy and safety of T-EUS procedures.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who has undergone clinically indicated and/or standard of care T-EUS procedures from October 2014 - May 2019
* Any patient who will undergo clinically indicated and/or standard of care T-EUS procedures from June 2019 - June 2027

Exclusion Criteria:

* Any patient who has not undergone endoscopic ultrasound would be excluded from the study.
* Below 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient who has undergone clinically indicated and/or standard of care T-EUS procedures
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-06-12 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
clinical success rates | October 2014 - June 2022
  Documentation of clinical success rates
Documentation of Safety | October 2014 - June 2022
  Number of subjects with Adverse Events; Type, frequency and intensity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Prashant Kedia, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided